CLINICAL TRIAL: NCT00200421
Title: A Double-Blind, Randomized, Multi-Center, Active Comparator, Five Treatment Study of the Effects of Nebivolol Compared to Atenolol on Cardiovascular Hemodynamics and Exercise Capacity in Patients With Mild to Moderate Hypertension
Brief Title: A Pilot Study Comparing Nebivolol and Atenolol and Its Effects With Exercise in Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Bertek Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEB203
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2003-08

CONDITIONS: Hypertension
Keywords: Nebivolol; Atenolol; Exercise; Hypertension
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Nebivolol; Atenolol

INTERVENTIONS:
Drug: Nebivolol and Atenolol

SUMMARY:
The purpose of this study is to determine the effects on exercise capacity of nebivolol compared to atenolol in hypertensive patients.

DETAILED DESCRIPTION:
This was a pilot, phase II, double-blind, randomized, muticenter, active-comparator, five treatment parallel group dosing and mechanistic study. The study consisted of two phases: 1) screen/washout/single-blind placebo run-in and 2) randomization/treatment. There was a minimum of five scheduled study visits.

ELIGIBILITY:
Inclusion Criteria:

* An average sitting diastolic blood pressure (DBP) of greater then or equal to 95 mmHg and less then or equal to 109 mmHg at baseline

Exclusion Criteria:

* Recent myocardial infarction or stroke
* Secondary Hypertension
* Contraindications to beta-blocker therapy or stopping prior antihypertensive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2002-05; Study Completion 2003-08

PRIMARY OUTCOMES:
The percent change in sub-maximal exercise duration by cycle ergometer at peak drug effect at end of treatment compared to baseline.

SECONDARY OUTCOMES:
The change in sub-maximal exercise duration at end of treatment compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Betty S. Riggs, MD, MBA, Study Director — Mylan Pharmaceuticals Inc
Locations (1):
- Mylan Pharmaceuticals Inc., Morgantown, West Virginia, United States